CLINICAL TRIAL: NCT06598735
Title: An Open, Multicenter Phase I Study of Safety, Tolerability, and Pharmacokinetics of HRS-4508 Monotherapy in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Clinical Study of the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of HRS-4508 Monotherapy in Patients With Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4508-101
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: monotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group: HRS-4508 (Experimental)
  Interventions: Drug: HRS-4508

INTERVENTIONS:
Drug: HRS-4508 — HRS-4508

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS-4508 in subjects with advanced or metastatic solid tumors and explore the reasonable dosage of HRS-4508.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing to participate in the study, sign the informed consent form, have good compliance, and cooperate with follow-up visits.
2. Aged 18-75 years, male or female.
3. Patients with advanced malignant tumors confirmed pathologically;
4. Failure of adequate standard treatment, or no effective standard treatment;
5. Patients must have at least 1 extracranial measurable target lesion per RECIST v1.1;
6. The expected survival period is more than 12 weeks;
7. The Eastern Cooperative Oncology Group (ECOG) physical fitness score is 0-1;
8. Have sufficient bone marrow and organ function (have not received blood transfusion or hematopoietic stimulating factor treatment within 14 days):

   ANC≥1.5 ×10e9/L; PLT≥100 × 10e9/L; Hb≥ 90 g/L; Cr）≤1.5 × times the upper limit of normal (ULN) or Clcr≥ 60 mL/min; LVEF≥50%; TBIL≤1.5 × times the upper limit of normal (ULN) ; ALT and AST ≤3×times the upper limit of normal (ULN)（Patients with liver metastasis, ≤5×ULN）; International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.
9. Female subjects of childbearing age must undergo a serum pregnancy test within 7 days before starting the study medication, and the result is negative, and are willing to use a medically approved high-efficiency contraception during the study period and within 1 months after the last administration of the study drug Measures.

Exclusion Criteria:

1. Subjects with a history of malignant tumors, except patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or cervical carcinoma in situ who have undergone possible curative treatment and did not have disease recurrence within 3 years since starting the treatment.
2. Subjects had cancerous meningitis or untreated central nervous system metastases.
3. Subjects had severe cardiovascular and cerebrovascular diseases.
4. There is third-space effusion that cannot be controlled by drainage and other methods (such as massive ascites, pleural effusion, pericardial effusion).
5. Subjects had or currently had idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug pneumonia, or CT during screening showed active pneumonia.
6. Arteriovenous thrombosis occurred within 6 months prior to the first dose.
7. Severe infection occurred within 4 weeks prior to initial administration.
8. Subjects with refractory nausea, vomiting, or other gastrointestinal disorders that affect the use of oral medications: including malabsorption syndrome.
9. Known history of human immunodeficiency virus (HIV) seropositive status or acquired immunodeficiency syndrome (AIDS).
10. Subjects had active hepatitis.
11. Subjects were scheduled to receive other systemic antitumor therapies during the study period.
12. Known allergies and contraindications to the investigational drug or any of its components.
13. Other factors as judged by the investigator that may lead to the termination of the study, such as other serious diseases, serious laboratory test abnormalities, or family or social factors that could affect the safety of the subject, or the collection of study data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints: Number of subjects with adverse events and the severity of adverse events | every 4 weeks after treatment initiation (through study completion, an average 5 mouths)
DLT (Dose-limiting toxicity) | during the first 21-day cycle of HRS-4508 treatment
MTD (Maximum tolerated dose) | 3 weeks after treatment initiation
RP2D (Recommended Phase II Dose) | 3 weeks after treatment initiation

SECONDARY OUTCOMES:
ORR (Objective response rate - RECIST 1.1) | Up to approximately 6 months
  ORR is defined as the proportion of subjects who have achieved complete response (CR) or partial response (PR) according to RECIST 1.1.
DoR (Duration of Response per RECIST 1.1) | Up to approximately 2 years
DCR (Disease control rate-RECIST 1.1) | Up to approximately 2 years
  DCR is defined as the proportion of subjects who have achieved stable disease(SD)、complete response (CR) or partial response (PR) according to RECIST 1.1.
PFS | Up to approximately 2 years
  Progression-free survival per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided